CLINICAL TRIAL: NCT07245199
Title: Protein Intake Distribution to Support Muscle Anabolism in Healthy Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL-010056 / METC25-038; NL-010056 / METC25-038 (Other: Maastricht University Medical Center)
Record Dates: First submitted 2025-10-02; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: No Condition, Healthy Individuals

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BALANCED (Experimental)
  Interventions: Dietary Supplement: protein intake
- SIP (Experimental)
  Interventions: Dietary Supplement: Protein intake
- BOLUS (Experimental)
  Interventions: Dietary Supplement: protein intake

INTERVENTIONS:
Dietary Supplement: protein intake — 1x 100g
  Arms: BOLUS
Dietary Supplement: protein intake — 4x 25 g
  Arms: BALANCED
Dietary Supplement: Protein intake — 15x 7 g
  Arms: SIP

SUMMARY:
The purpose of the study is to evaluate whether the distribution pattern of daily protein intake affects how much muscle protein can be built in the muscle after resistance exercise and at rest.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-40 years
* Healthy
* 18.5 ≤ BMI 30 ≤ kg・m-2

Exclusion Criteria:

* Smoking
* Sports/exercise >4 sessions/week or a structured resistance or endurance training schedule
* Lactose intolerant or allergies to milk protein
* A history of neuromuscular problems
* Use of anticoagulation medication
* Individuals on any medications known to affect protein metabolism (i.e. , non-steroidal anti-inflammatories, or prescription acne medications).
* Strict vegetarian
* Injury or condition that would limit the participant from performing the resistance exercise.
* Pregnancy
* Hormone replacement therapy
* Blood donation within the past 2 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
fractional synthetic rate | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Result] Mamerow MM, Mettler JA, English KL, Casperson SL, Arentson-Lantz E, Sheffield-Moore M, Layman DK, Paddon-Jones D. Dietary protein distribution positively influences 24-h muscle protein synthesis in healthy adults. J Nutr. 2014 Jun;144(6):876-80. doi: 10.3945/jn.113.185280. Epub 2014 Jan 29. PMID 24477298
- [Result] Areta JL, Burke LM, Ross ML, Camera DM, West DW, Broad EM, Jeacocke NA, Moore DR, Stellingwerff T, Phillips SM, Hawley JA, Coffey VG. Timing and distribution of protein ingestion during prolonged recovery from resistance exercise alters myofibrillar protein synthesis. J Physiol. 2013 May 1;591(9):2319-31. doi: 10.1113/jphysiol.2012.244897. Epub 2013 Mar 4. PMID 23459753